CLINICAL TRIAL: NCT03049982
Title: A Study for Obstructive Sleep Apnea Using a New At-Home Sleep Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zephyr Sleep Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZCP2016_03
Record Dates: First submitted 2017-02-06; First posted 2017-02-10 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Oral appliance therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMP test group (Other): All individuals will undergo a test using the auto-titrating mandibular positioner.
  Interventions: Device: Auto-titrating mandibular positioner test

INTERVENTIONS:
Device: Auto-titrating mandibular positioner test — Participants will undergo a theragnostic test using the auto-titrating mandibular positioner to determine if they are eligible candidates to use oral appliance therapy for their obstructive sleep apnea. The device works by moving the lower jaw forward in response to respiratory events while the participant sleeps. All participants will undergo the same test.

SUMMARY:
The purpose of the study is to test the workflow of an auto-titrating mandibular positioner in its intended setting. Participants with obstructive sleep apnea will use the device to determine their eligibility for oral appliance therapy and provide feedback on usability of the device.

DETAILED DESCRIPTION:
One treatment for obstructive sleep apnea is oral appliance therapy during sleep, in which an appliance that covers the upper and lower teeth acts to pull the lower jaw forward, opening the throat passage and allowing for normal breathing. However, oral appliance therapy does not treat sleep apnea effectively in all individuals. In order to identify those individuals for whom oral appliance therapy will work, the study sponsor has developed an investigational device called an auto-titrating mandibular positioner.

The device automatically pulls the lower jaw forward in response to respiratory events while the individual sleeps. Study participants will learn the outcome of their sleep tests and will provide feedback on the ease of use of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 18 years of age
2. Participant has been deemed suitable for oral appliance therapy
3. Prescription for oral appliance
4. Adequate range of motion
5. Adequate dentition
6. Ability to understand and provide informed consent
7. Ability and willingness to meet the required schedule

Exclusion Criteria:

1. Loose teeth or advanced periodontal disease
2. Full dentures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Integration of the device into the existing workflow of a dental sleep medicine practice | 6 months
  Data for this outcome are largely directed at the study staff, not study participants. Data collected for this outcome include: time required to evaluate eligibility for device use, time required to prepare device for use.
Convenience/feasibility of carrying out a multi-night AMP study in the home | 6 months
  Participants will complete a questionnaire following their AMP tests to collect data on participants' opinion of the device (includes opinion of various device components, ease of use of the device).
Feasibility of instructing the participant on the use of the AMP device at the practitioner's office | 6 months
  Data for this outcome are directed at study staff, not study participants. Data collected will include feedback on ease of training participants on device use. Participants will be asked if they felt they received adequate training from the study staff via a questionnaire.

SECONDARY OUTCOMES:
Time to therapy | 6 months
  Time to therapy will be evaluated by tracking the time from the first consultation at the dentist's office to the setting of the temporary appliance (for individuals whose tests indicate they are predicted candidates for oral appliance therapy).
Number of study visits | 6 months
  The number of study visits will be recorded. This data will be collected from study records and does not require input from the participant.
Length of study visits | 6 months
  The length of each visit (minutes) will be recorded. This data will be collected from study records and does not require input from the participant.
Ease of scheduling study visits | 6 months
  The ease of scheduling will be discussed with the study staff to collect data on ease of integration of the device into the practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Encino Center for Sleep and TMJ Disorders, Encino, California, United States

IPD SHARING:
Plan to Share IPD: No